CLINICAL TRIAL: NCT07155798
Title: Eco-friendly or Effective? Evaluating Plaque Removal in Adolescents Using Bamboo and Conventional Plastic Toothbrushes: a Randomized Controlled Trial
Brief Title: Evaluating Plaque Removal in Adolescents Using Bamboo and Conventional Plastic Toothbrushes
Acronym: prevention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heba Helal (Other)
Responsible Party: Sponsor-Investigator, Heba Helal, lecturer, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CU5-6-2025
Record Dates: First submitted 2025-05-06; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Plaque Removal
Keywords: bamboo; conventional toothbrush; plaque removal

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- conventional toothbrush (Active Comparator): conventional toothbrush
  Interventions: Device: bamboo toothbrush; Device: conventional toothbrush
- bamboo toothbrush (Experimental): recent tooth brush
  Interventions: Device: bamboo toothbrush; Device: conventional toothbrush

INTERVENTIONS:
Device: bamboo toothbrush — recent toothbrush
  Other Names: charcoal toothbrush
Device: conventional toothbrush — conventional toothbrush

SUMMARY:
evaluation of bamboo and conventional toothbrushes in plaque removal

DETAILED DESCRIPTION:
evaluation of the use of two tooth brushed bamboo and conventional tooth brushes in plaque removal in adolescence

ELIGIBILITY:
Inclusion Criteria: healthy and medically free participants

-

Exclusion Criteria:

* disabled participants who cannot perform tooth brushing

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
plaque score | T0 baseline, T1 at 7 days and T2 at 2 weeks
  measurement of plaque accumulation in scale from 0 till 5 0 indicates no plaque and 5 indicated 2/3 of the tooth surface is covered with plaque

SECONDARY OUTCOMES:
bristle contamination | after 2 weeks
  bacterial count on toothbrush bristle

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt